CLINICAL TRIAL: NCT02591953
Title: Prospective Clinical Analysis of Ultrasound-guided Biceps Corticosteroid Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to meet enrollment and follow up criteria
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jeremy A Alland, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15101504
Record Dates: First submitted 2015-10-21; First posted 2015-10-30 (Estimated); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Biceps Tendonitis; Injection
MeSH Terms: interventions — Methylprednisolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Ultrasound-guided Injection (Experimental): Injection performed with ultrasound-guidance
  Interventions: Procedure: Ultrasound-guidance; Drug: Methylprednisolone; Drug: Lidocaine 1%
- Landmark-guided Injection (Active Comparator): Injection performed at point of maximal tenderness along biceps tendon
  Interventions: Procedure: Landmark-guidance; Drug: Methylprednisolone; Drug: Lidocaine 1%

INTERVENTIONS:
Procedure: Ultrasound-guidance — Using ultrasound-guidance to perform a corticosteroid injection
  Arms: Ultrasound-guided Injection
Procedure: Landmark-guidance — Using landmark-guidance to perform a corticosteroid injection
  Arms: Landmark-guided Injection
Drug: Methylprednisolone — Corticosteroid used in injection (40 mg)
Drug: Lidocaine 1% — Anesthesic used in injection

SUMMARY:
Using randomization, prospectively determine superiority of either ultrasound-guided or landmark-guided biceps corticosteroid injections with regard to various clinical variables.

DETAILED DESCRIPTION:
Patients are diagnosed with biceps tendinitis in the outpatient clinic. After diagnosis, all the patients that meet inclusion/exclusion criteria will be offered to enroll in the study. Study will be described to the patient with regard to protocol and consent. All questions regarding the study will be answered, and it will be explicitly described that the study involvement will not change clinical care. It will be explained that investigators expect a follow up appointment at minimum at three weeks and three months. There may be further follow up requested up to 1 year from enrollment.

After collection of informed consent, the patient will be randomized to either ultrasound-guided or landmark-guided injection. The patient will complete clinical scores at the initial visit prior to the injection. After injection, the patient will have follow up scheduled for three weeks and three months. To ensure patient blinding, an ultrasound will be placed on the patient for both groups, but only active imaging with be performed for the ultrasound-guided patient group. For clinician blinding, a different clinician than the injecting clinician will perform the follow up examinations. The patient is instructed to not seek additional injections or physical therapy during the study.

ELIGIBILITY:
Inclusion Criteria:

* Pain at intertubercular groove
* Anterior humeral pain
* Positive Speed's Test
* Bicep's tendinitis is primary diagnosis for patient
* Patient agrees to follow up and consent

Exclusion Criteria:

* Prior biceps surgery or injections
* Prior SLAP or labral repair
* Concomitant shoulder arthroplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Orthopeadics at Rush, Chicago, Illinois, United States

REFERENCES:
- [Background] Hashiuchi T, Sakurai G, Morimoto M, Komei T, Takakura Y, Tanaka Y. Accuracy of the biceps tendon sheath injection: ultrasound-guided or unguided injection? A randomized controlled trial. J Shoulder Elbow Surg. 2011 Oct;20(7):1069-73. doi: 10.1016/j.jse.2011.04.004. Epub 2011 Jul 22. PMID 21782470
- [Background] Zhang J, Ebraheim N, Lause GE. Ultrasound-guided injection for the biceps brachii tendinitis: results and experience. Ultrasound Med Biol. 2011 May;37(5):729-33. doi: 10.1016/j.ultrasmedbio.2011.02.014. Epub 2011 Mar 31. PMID 21458143
- [Background] Ucuncu F, Capkin E, Karkucak M, Ozden G, Cakirbay H, Tosun M, Guler M. A comparison of the effectiveness of landmark-guided injections and ultrasonography guided injections for shoulder pain. Clin J Pain. 2009 Nov-Dec;25(9):786-9. doi: 10.1097/AJP.0b013e3181acb0e4. PMID 19851159
- [Background] Naredo E, Cabero F, Beneyto P, Cruz A, Mondejar B, Uson J, Palop MJ, Crespo M. A randomized comparative study of short term response to blind injection versus sonographic-guided injection of local corticosteroids in patients with painful shoulder. J Rheumatol. 2004 Feb;31(2):308-14. PMID 14760802
- [Background] Aly AR, Rajasekaran S, Ashworth N. Ultrasound-guided shoulder girdle injections are more accurate and more effective than landmark-guided injections: a systematic review and meta-analysis. Br J Sports Med. 2015 Aug;49(16):1042-9. doi: 10.1136/bjsports-2014-093573. Epub 2014 Nov 17. PMID 25403682
- See also: AMSSM Statement of Interventional Musculoskeletal Ultrasound — http://journals.lww.com/cjsportsmed/Fulltext/2015/01000/American_Medical_Society_for_Sports_Medicine.2.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound-guided Injection | Landmark-guided Injection
Started | 12 | 10
Completed | 6 | 4
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound-guided Injection | Landmark-guided Injection | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 10 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
Pain and Function Scores [Mean (Standard Deviation); unit: units on a scale] — VAS
  units on a scale | NA (NA) — Data was not analyzed and was lost when PRO company changed | NA (NA) — Data was not analyzed and was lost when PRO company changed | NA (NA) — Data was not analyzed and was lost when PRO company changed

OUTCOME MEASURES:

1. Primary Outcome: Simple Shoulder Test
Description: 12 question assessment of shoulder function with yes or no answers
Time Frame: 1 year
Population: The study was terminated and data could not be analyzed as the department switched PRO companies. Access to the data was lost at that time.
Groups:
- Results: Results not reported
Arm/Group | Results
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year after injection
Arm/Group | Ultrasound-guided Injection | Landmark-guided Injection
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-03-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT02591953/Prot_000.pdf